CLINICAL TRIAL: NCT02803697
Title: Predictive Factors of Recurrence of Non Functioning Pituitary Adenomas : a Retrospective Study of 220 Patients in the Reims University Hospital, France
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA13045
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pituitary Adenomas
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients: All patients who underwent surgery for a NFPA in Reims university hospital between 01/01/1991 and 31/12/2004
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients

SUMMARY:
Non functioning pituitary adenomas (NFPAs) are the most common pituitary adenomas. Their growth is usually slow and diagnosis is often made in the context of masse effect .The therapeutic alternatives are surgery and radiotherapy such as fractionated stereotactic radiotherapy. Nowadays, there is no clinical or histological prognostic factor to allow an individualized follow-up and recurrence could happen 10 or 15 years after the first surgery. In this study, the investigators evaluate NFPAs recurrence rate after surgery and try to find predictive factors of recurrence to personalized the follow-up of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year-old
* diagnosis of NFPAs confirmed with hormonal and histological analysis
* patients who underwent surgery in neurosurgery unit of the Reims university hospital between 01/01/1991 and 31/12/2004

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgery for a NFPA in Reims university hospital between 01/01/1991 and 31/12/2004, at least 10 years of follow-up. One group.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate / predictive factors of recurrence | up to 21 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France